CLINICAL TRIAL: NCT04522687
Title: Observation of the Impact of Radiotherapy With or Without Chemotherapy in the Value of Peripheral Blood Lymphocyte Subsets for Patients With Thoracic Cancer
Brief Title: Influence of Radiotherapy and Chemotherapy in the Value of Peripheral Blood Lymphocyte Subsets Among Thoracic Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Cancer Hospital, China (Other)
Responsible Party: Principal Investigator, Fan Min, MD. PhD, Shanghai Cancer Hospital, China
Other Study IDs: SHCH1501
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: NSCLC; Esophageal Squamous Cell Carcinoma; Thymic Epithelial Tumor
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Thymic epithelial tumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observation, single center study to evaluate the alternations and prognostic value of peripheral blood lymphocyte (PBL) in patients diagnosed with thoracic cancers, including lung cancer, esophageal squamous cell carcinoma and thymic epithelial carcinoma underwent radiotherapy with or without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Age at least 18 years. ECOG PS 0-1. Pathologically confirmed NSCLC, esophageal squamous cell carcinoma or thymic epithelial tumor.

Life expectancy of more than 3 months. Patients with no indications for palliative radiotherapy in the opinion of the investigator.

Patients with a prior history of surgery are eligible if they have recovered adequately from the toxicity and/or complications of surgery.

Signed informed consent for the use of fresh tumor biopsies before and during the treatment.

Women of childbearing age and men must agree to use effective contraception during the trial.

Adequate organ function within 1 week prior to the enrollment：

1. Adequate bone marrow function: hemoglobin ≥80g/L, white blood cell (WBC) count ≥ 4.0 * 10 ^ 9/L or neutrophil count ≥ 1.5 * 10 ^ 9/L, and platelet count ≥ 100 * 10 ^ 9/L;
2. Adequate hepatic function: total bilirubin < 1.5 x upper limit of normal (ULN). Note: If total bilirubin is > 1.5 x ULN, direct bilirubin must ≤ ULN, Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤2.5 ULN;
3. Adequate renal function: serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min;

Exclusion Criteria:

Pregnant or lactating women. History of any other malignancy. Patients in whom palliative radiotherapy is indicated in the opinion of the investigator.

Active infection, congestive heart failure, myocardial infarction within the 6 months prior to enrollment, unstable angina pectoris or cardiac arrhythmia.

Patients who have received tumor vaccine; or administration of live, attenuated vaccine within 4 weeks before the start of treatment.

Mental disorders, drug abuse, and social condition that may negatively impact compliance in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients diagnosed with NSCLC, esophageal squamous cell carcinoma or thymic epithelial tumor.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Five years
  OS was defined as the time from the date of enrollment until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.

SECONDARY OUTCOMES:
Progression Free Survival | Five years
  PFS was measured from the date of enrollment to the date of disease progression as defined by Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 or death due to any cause, whichever occurred first

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China